CLINICAL TRIAL: NCT00302302
Title: The Effects of Increasing Doses of L-arabinose in a Sucrose Rich Meal on Intestinal Sucrase Activity in Man
Brief Title: The Effects of L-arabinose on Intestinal Sucrase Activity in Man
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Danisco (Industry)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: (KF) 01 270121; M181
Record Dates: First submitted 2005-09-21; First posted 2006-03-14 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Blood Glucose
Keywords: Blood glucose; Insulin; Triglyceride; GIP; GLP-1; L-arabinose; Appetite; Energy intake
MeSH Terms: conditions — Insulin Resistance | interventions — Arabinose

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: L-arabinose

SUMMARY:
The purpose of this study is to investigate the effect of L-arabinose in a sugar-rich meal on intestinal sucrase activity in healthy volunteers by measuring postprandial blood glucose and insulin, and selected intestinal hormonal responses to increasing doses of L-arabinose.

DETAILED DESCRIPTION:
Background:

The intake of common table sugar (sucrose) in the industrialised countries is relatively high. In Denmark the daily intake of sugar is in the range of 30-40 g/d exclusive the intake of sugar containing drinks. The health consequences of this relatively high sugar intake are heavily debated in the media. One of the arguments is that a high sugar intake may be one of the factors involved in the development of the metabolic syndrome, including overweight, increased blood glucose and insulin levels as well as impaired insulin action.

L-arabinose is widely distributed in plants and is a common component in plant cell walls in maize, wheat, rye, rice, plant gums etc. The isolated 5-carbon sugar has been shown to suppress the increase of blood glucose and plasma insulin after ingestion of sucrose in rats by inhibition of sucrase activity. In vitro studies on Caco-2 cells indicate that L-arabinose is a potent inhibitor on sucrase activity, possibly in a non-competitive way.

Potential nutritional advantages of consuming L-arabinose in combination with sucrose may therefore be a delayed digestion of sucrose and a lower absorption of glucose, resulting in both lower blood glucose and insulin levels. A delayed digestion of sucrose will reduce the energy utilisation with the potential of reducing weight gain in human subjects.

Methods:

This dose-response study with 14 healthy male volunteers has a randomised cross-over design based on four single "meals" separated by one week wash-out periods. Sugar rich drinks supplemented with different doses of L-arabinose will be tested with respect to postprandial blood glucose, insulin, triglyceride, glucose-dependent insulinotropic peptide (GIP) and glucagon-like peptide-1 (GLP-1). Postprandial blood samples will be taken every 15 to 30 min for 180 min. Appetite sensations will be measured every 30 min during the experiment. After 180 minutes a lunch will be served and energy intake (EI) will be registered.

ELIGIBILITY:
Inclusion Criteria:

* healthy males
* BMI between 18.4-25 kg/m2
* age between 18 and 30

Exclusion Criteria:

* donation of blood 3 months before or during the study
* gastrointestinal disorders, diabetes, hypertension, hyperlipidemia, chronic infectious disease (HIV or hepatitis)
* smoking
* consumption of more than 21 alcoholic drinks/week
* elite athletes
* on medication

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-09; Primary Completion 2005-11 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Plasma glucose, insulin, triglycerides, GIP and GLP-1 | 2 hours
  Blood samples 2 hours after a test meal

SECONDARY OUTCOMES:
Appetite measurements and energy intake | 10 hours
  measured after a test meal

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Bukhave, MSc, MScD, Principal Investigator — Institute of Human Nutrition, The Royal Veterinary and Agricultural University, Denmark
Locations (1):
- Institute of Human Nutrition, The Royal Veterinary and Agricultural University, Frederiksberg, Denmark

REFERENCES:
- [Derived] Krog-Mikkelsen I, Hels O, Tetens I, Holst JJ, Andersen JR, Bukhave K. The effects of L-arabinose on intestinal sucrase activity: dose-response studies in vitro and in humans. Am J Clin Nutr. 2011 Aug;94(2):472-8. doi: 10.3945/ajcn.111.014225. Epub 2011 Jun 15. PMID 21677059